CLINICAL TRIAL: NCT02643108
Title: Randomized Controlled Clinical Trial of Lateral Episiotomy Versus no Episiotomy in Vacuum Assisted Delivery in Non-parous Women
Brief Title: Lateral Episiotomy or Not in Vacuum Assisted Delivery in Non-parous Women
Acronym: EVA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Sophia Brismar Wendel, MD, PhD, Dept of Women's health, Danderyd Hospital, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015/1238-31/2
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Floor Disorders; Fecal Incontinence; Dystocia; Fetal Hypoxia
Keywords: Lateral episiotomy; Obstetric anal sphincter injury; Vacuum extraction; Anal incontinence
MeSH Terms: conditions — Pelvic Floor Disorders; Fecal Incontinence; Dystocia; Fetal Hypoxia; Encopresis

STUDY DESIGN:
Masking Description: The allocation will be masked during statistical analyses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lateral episiotomy (Experimental): Lateral episiotomy (left or right) is performed by the attending physician or assisting midwife at crowning of the fetal head in operative vaginal delivery by vacuum extraction. Regular manual perineal support is applied.
  Interventions: Procedure: Lateral episiotomy
- No episiotomy (No Intervention): No episiotomy is performed during operative vaginal delivery, unless vitally indicated (for example severe fetal distress). The woman may tear spontaneously. Regular manual perineal support is applied.

INTERVENTIONS:
Procedure: Lateral episiotomy — When the woman is randomized to episiotomy, lateral episiotomy is performed with scissors on the left or right side of the vaginal opening. Origin of incision is 1.0 - 3.0 cm from the midline/posterior forchette and is cut 3.0 cm or more towards the ischial tuberosity at an angle of 60 degrees from the midline.
  Arms: Lateral episiotomy

SUMMARY:
Nulliparous women with a live singleton pregnancy in cephalic presentation past 34 gestational weeks will be randomized to lateral episiotomy or no episiotomy when operative vaginal delivery by vacuum extraction is indicated. Primary outcome is clinically diagnosed obstetric anal sphincter injury (OASIS) of any degree.

DETAILED DESCRIPTION:
The study started at Danderyd Hospital 30 June 2017. Danderyd Hospital is a large teaching hospital affiliated to Karolinska Institutet in Stockholm, Sweden. South General Hospital in Stockholm, Uppsala University Hospital, Falun Hospital, Helsingborg Hospital, Växjö Hospital, Umeå University Hospital, and Gothenburg University Hospital Östra have joined the trial 2017-2019. The trial had included 717 women of planned 710 women by 15 February 2023.

Informed consent was collected from nulliparous women with a singelton, live fetus in cephalic presentation, with a planned vaginal delivery and without previous gynecological surgery for incontinence or genital prolapse. Women were approached at any time from gestational week 18 until delivery, unless they were in severe pain or discomfort, or there was not enough time to consider the information, or any other reason not to obtain consent. The informed consent forms are kept at the receiving research department and a note of consent/no consent was made in the obstetric medical record.

At indication for vacuum extraction, the patient's consent was confirmed verbally and allocation was made via sealed opaque envelopes on the vacuum extraction equipment mobile cart. Randomization was performed 1:1 in random permuted blocks generated electronically by an external organization (Karolinska Trial Alliance).

Lateral episiotomy was performed according to the intervention description. A reduction of OASIS from 12.4% to 6.2% can be detected with 80% power and less than 5% risk of alpha-error (p<0.05) with 355 women in each group using Chi-square test comparing two independent proportions in a two-sided test (3% missing outcome). A smaller reduction is clinically valuable, although the risk-benefit relationship between receiving a prophylactic episiotomy and the chance of an intact perineum may limit the feasibility of a larger trial in a setting with a restrictive episiotomy policy. We have obtained ethical approval to randomise a total of 1400 women, which enables us to detect a reduction in OASIS rate at VE from 12.4% to 7.8% (p<0.05). We planned and performed an interim analysis in order to exclude an unethically large difference (p<0.01) at 350 randomised women. The stopping criteria were not met. In 2019, we decided to aim for 710 randomised women due to slow recruitment.

Data was collected prospectively through Case Record Forms and the obstetric medical record Obstetrix (Cerner Sverige AB), which covers approximately 98% of deliveries with complete data, and the Swedish Pregnancy Register covering 98% of births in Sweden from 2015. Using a weblink, questionnaires from the national Obstetric Perineal Tear Register, are sent out electronically for the follow-up of study participants. In addition, questionnaires regarding birth satisfaction/experience (BSS-R and CEQ 2.0) are sent at 8 weeks after delivery. Questionnaires regarding sexual function (FSFI and FSDS) and quality of life (Euro-QoL-5D) at delivery and after 12 months.

A follow-up from registers regarding mode of delivery and prevalence of episiotomy and OASIS in subsequent births will be performed at 5 years and 10 years after the index birth.

A substudy takes place in Stockholm, Uppsala, and Helsingborg, where randomised women are examined at 6-12 months after delivery with 3D endovaginal and endoanal ultrasound to detect levator and sphincter injuries, measure episiotomy scars, establish POP-Q scores, and evaluate a new questionnaire for pelvic floor function after perineal tears.

Another substudy has taken place in Stockholm and Falun, where women who have been asked for consent (both affirmative and non-affirmative responders), as well as midwives who have tried to obtain consent, were invited to a qualitative interview study to explore the recruitment experience of women and midwives.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women,18 years old or more, able to give written informed consent in Swedish or English, with a live singleton pregnancy, in a cephalic presentation over 34 completed gestational weeks with a medical indication for vacuum extraction.

Exclusion Criteria:

* Previous vaginal or perineal surgery for incontinence or genital prolapse, any contra-indication to vacuum extraction (ie fetal disorder or malformation).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 717 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Obstetric anal sphincter injury | 1 hour
  Rupture or tear of the external and/or internal anal sphincter at any degree (third and fourth degree perineal tear); International Classification of Diseases (ICD)-10 O70.2 or O70.3.

SECONDARY OUTCOMES:
Other degree of perineal or vaginal tear | 1 hour
  Rupture, tear or hematoma in the perineum or vagina; International Classification of Diseases (ICD)-10 O70.0, O70.1, O70.9, O71.4-9.
Maternal blood loss at delivery | 6 hours
  Estimated blood loss in milliliters through weighing of sheets and drapes during and up to 6 hours after delivery.
Neonatal scalp injury | 24 hours
  Prevalence (number of patients) of scalp injury to the neonate after instrumental delivery, such as open wounds, cephalic hematoma, subgaleal hematoma, and intracranial hemorrhage, according to diagnose by neonatologist.
Pain experience | 1 day, 8 weeks, 1 year
  Numeric Rating Scale (0-10, where 0 is no pain and 10 is worst possible pain) estimated pain through questionnaire at baseline (first days post partum), 8 weeks and 12 months after delivery and at 8 weeks through questionnaires: number of days using analgetic medication.
Birthing experience | 1 day, 8 weeks
  Numeric Rating Scale (1-10, where 1 is worst possible experience and 10 is best possible experience) 1-7 days postpartum, Questionnaire at 8 weeks after delivery regarding patient satisfaction using the Birth Satisfaction Scale Revised (short form) and the Childbirth Experience Questionnaire 2.0.
Anal incontinence | 8 weeks, 1 year, and 5 years
  Questionnaire at baseline, 8 weeks, 1 year, and 5 years after delivery through the Swedish Perineal Laceration Register regarding anal continence function (Wexner score based).
Sexual function | 1 year and 5 years
  Questionnaire at baseline (first day post partum), 1 year, and 5 years after delivery through the Swedish Obstetrical Tear Register, as well as the Female Sexual Function Index and Female Sexual Distress Score Questionnaires.
Pelvic organ prolapse symptoms | 1 year and 5 years
  Questionnaire at baseline, 1 year, and 5 years after delivery through the Swedish Perineal Laceration Register regarding symptoms of pelvic organ prolapse.
Quality of life score | 1 year and 5 years
  Assessment of quality of life by questionnaire at baseline, 1 year, and 5 years using the Euro-QoL-5D.
Mode of delivery in subsequent birth | 5 years and 10 years
  Register data will be extracted from the Swedish Pregnancy Register.
Prevalence of obstetric anal sphincter injury in subsequent birth | 5 years and 10 years
  Register data will be extracted from the Swedish Pregnancy Register.
Prevalence of episiotomy in subsequent birth | 5 years and 10 years
  Register data will be extracted from the Swedish Pregnancy Register.

CONTACTS AND LOCATIONS:
Overall Officials: Sophia Brismar Wendel, MD, PhD, Principal Investigator — Karolinska Institutet Danderyd Hospital
Locations (8):
- Sweden (8):
  - Falun Hospital, Falun
  - Östra Hospital Gothenburg University, Gothenburg
  - Helsingborg Hospital, Helsingborg
  - Danderyd Hospital, Stockholm
  - South General Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala
  - Växjö Hospital, Vaxjo

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data on the primary outcome will be shared with other researchers for a joint publication.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When results have been published (after 1 year).
Access Criteria: Anonymized data on the primary outcome will be shared with other researchers for a joint publication.

REFERENCES:
- [Background] Laine K, Pirhonen T, Rolland R, Pirhonen J. Decreasing the incidence of anal sphincter tears during delivery. Obstet Gynecol. 2008 May;111(5):1053-7. doi: 10.1097/AOG.0b013e31816c4402. PMID 18448735
- [Background] Murphy DJ, Macleod M, Bahl R, Goyder K, Howarth L, Strachan B. A randomised controlled trial of routine versus restrictive use of episiotomy at operative vaginal delivery: a multicentre pilot study. BJOG. 2008 Dec;115(13):1695-702; discussion 1702-3. doi: 10.1111/j.1471-0528.2008.01960.x. PMID 19035944
- [Background] Kalis V, Laine K, de Leeuw JW, Ismail KM, Tincello DG. Classification of episiotomy: towards a standardisation of terminology. BJOG. 2012 Apr;119(5):522-6. doi: 10.1111/j.1471-0528.2011.03268.x. Epub 2012 Feb 3. PMID 22304364
- [Background] de Leeuw JW, de Wit C, Kuijken JP, Bruinse HW. Mediolateral episiotomy reduces the risk for anal sphincter injury during operative vaginal delivery. BJOG. 2008 Jan;115(1):104-8. doi: 10.1111/j.1471-0528.2007.01554.x. Epub 2007 Nov 12. PMID 17999693
- [Background] Raisanen SH, Vehvilainen-Julkunen K, Gissler M, Heinonen S. Lateral episiotomy protects primiparous but not multiparous women from obstetric anal sphincter rupture. Acta Obstet Gynecol Scand. 2009;88(12):1365-72. doi: 10.3109/00016340903295626. PMID 19852569
- [Derived] Bergendahl S, Jonsson M, Hesselman S, Ankarcrona V, Leijonhufvud A, Wihlback AC, Wallstrom T, Rydstrom E, Friberg H, Kopp Kallner H, Brismar Wendel S. Lateral episiotomy or no episiotomy in vacuum assisted delivery in nulliparous women (EVA): multicentre, open label, randomised controlled trial. BMJ. 2024 Jun 17;385:e079014. doi: 10.1136/bmj-2023-079014. PMID 38886011
- [Derived] Ericson J, Anagrius C, Rygaard A, Guntram L, Wendel SB, Hesselman S. Women's experiences of receiving information about and consenting or declining to participate in a randomized controlled trial involving episiotomy in vacuum-assisted delivery: a qualitative study. Trials. 2021 Sep 26;22(1):658. doi: 10.1186/s13063-021-05624-8. PMID 34565424
- [Derived] Bergendahl S, Ankarcrona V, Leijonhufvud A, Hesselman S, Karlstrom S, Kopp Kallner H, Brismar Wendel S. Lateral episiotomy versus no episiotomy to reduce obstetric anal sphincter injury in vacuum-assisted delivery in nulliparous women: study protocol on a randomised controlled trial. BMJ Open. 2019 Mar 13;9(3):e025050. doi: 10.1136/bmjopen-2018-025050. PMID 30872546
- See also: University based site for the trial (in Swedish) — https://ki.se/kids/eva-studien
- See also: Swedish Network for National Clinical Studies in Obstetrics and Gynecology — https://www.snaks.se/en/start/

DOCUMENTS (1):
  • Study Protocol (2019-04-18): https://cdn.clinicaltrials.gov/large-docs/08/NCT02643108/Prot_000.pdf